CLINICAL TRIAL: NCT05319353
Title: A Phase 3, Open-label, Single-arm, Repeated-dose Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Antiviral Activity of Maribavir for the Treatment of Cytomegalovirus (CMV) Infection in Children and Adolescents Who Have Received a Hematopoietic Stem Cell Transplant (HSCT) or a Solid Organ Transplant (SOT)
Brief Title: A Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Antiviral Activity of Maribavir for the Treatment of Cytomegalovirus (CMV) Infection in Children and Adolescents Who Have Received a Hematopoietic Stem Cell Transplant (HSCT) or a Solid Organ Transplant (SOT)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-2004; 2021-004279-15 (EudraCT Number); jRCT2031230753 (Registry Identifier: jRCT); 2023-508988-73-00 (EU CTIS Number: EU Trial Number)
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cytomegalovirus (CMV)
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Intervention Model Description: Three dosing cohorts based on participant's age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Maribavir 400, 200 or 100 mg (Experimental): Participants with greater than or equal to (>=) 12 to less than (<) 18 years of age will receive maribavir 400 milligrams (mg) (2*200 mg tablets or powder for oral suspension) twice daily (BID) based on body weight >= 25 kilogram (kg); or 200 mg tablet or powder for oral suspension BID based on body weight 14 to < 25 kg; or 100 mg powder for oral suspension BID based on body weight 10 to < 14 kg for up to 8 weeks treatment period (Day 1/Week 0 to Day 56/Week 8).
  Interventions: Drug: Maribavir
- Cohort 2: Maribavir 400, 200 or 100 mg (Experimental): Participants with >= 6 to < 12 years of age will receive maribavir 400 mg (2*200 mg tablets or powder for oral suspension) BID based on body weight >= 25 kg; or 200 mg tablet or powder for oral suspension BID based on body weight 14 to < 25 kg; or 100 mg powder for oral suspension BID based on body weight 10 to < 14 kg orally for up to 8 weeks treatment period (Day 1/Week 0 to Day 56/Week 8).
  Interventions: Drug: Maribavir
- Cohort 3: Maribavir 400, 200, 100 or 50 mg (Experimental): Participants with 0 to < 6 years of age will receive maribavir 400 mg (2*200 mg tablets or powder for oral suspension) BID based on body weight >= 25 kg; or 200 mg tablet or powder for oral suspension BID based on body weight 14 to < 25 kg; or 100 mg powder for oral suspension BID based on body weight 10 to < 14 kg; or 50 mg powder for oral suspension BID based on body weight 7 to < 10 kg; or 50 mg powder for oral suspension once daily (QD) based on body weight 5 to <7 kg for up to 8 weeks treatment period (Day 1/Week 0 to Day 56/Week 8).
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Participants will receive maribavir.
  Other Names: TAK-620

SUMMARY:
The main aim of this study is to find out the safety, tolerability and pharmacokinetics (PK) of maribavir for the treatment of CMV infection in children and teenagers after HSCT or SOT and to identify the optimal dose of maribavir using a 200 milligrams (mg) tablet formulation or powder for oral suspension.

The participants will be treated with maribavir for 8 weeks.

Participants need to visit their doctor during 12-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Parent/both parents or legally authorized representative (LAR) must provide signature of informed consent and there must be documentation of assent by the participant, as age appropriate, before completing any study-related procedures.
* Be a male or female child or adolescent < 18 years of age at the time of consent. For participants in Cohort 3 only (0 to <6 years) must have a gestational age of at least 39 weeks and a minimum weight of 5 kg.
* Be a recipient of an SOT or an HSCT that is functioning at the time of screening.
* Have a documented CMV infection which may be a first episode of post-transplant CMV viremia (primary or reactivation) or refractory to other anti-CMV treatments, with a CMV DNA screening value of >= 1365 International Units per milliliter (IU/mL) in whole blood or >= 455 IU/mL in plasma in 2 consecutive assessments separated by at least 1 day, as determined by local laboratory quantitative polymerase chain reaction (qPCR) or comparable quantitative nucleic acid amplification test (qNAAT) results. Quantitative assays must be standardized to the World Health Organization (WHO) CMV International Standard. Both samples must be taken within 14 days of first dose of study drug, with the second sample obtained within 5 days prior to first dose of study drug. The same laboratory and same sample type (whole blood or plasma) must be used for both assessments. If documented and verified values are available in medical history that fulfill this criterion entirely, they may be used instead.
* Have all the following results as part of screening laboratory assessments:
* Absolute neutrophil count >= 500 per cubic millimeter (/mm^3) (0.5 × 10^9 per liter [/L])
* Platelet count >= 15,000/mm^3 (15 × 10^9/L)
* Hemoglobin >= 8 grams per deciliter (g/dL) (>=80 grams per liter [g/L]).
* Have an estimated glomerular filtration rate (creatinine-based Bedside Schwartz equation) >= 30 milliliters per minute (mL/min) /1.73 meter square (m^2).
* Be a female of nonchildbearing potential. If a female of childbearing potential, have a negative serum human chorionic gonadotropin (hCG) or beta-human chorionic gonadotropin (β-hCG) pregnancy test at screening. Males, or nonpregnant, nonlactating females who are sexually active must agree to comply with the applicable contraceptive requirements of this protocol during the study treatment administration period and for 90 days after the last dose of study treatment.
* Have life expectancy of >= 8 weeks.
* Be willing and have an understanding and ability to fully comply with the study procedures and restrictions defined in the protocol. For younger children, the parent/both parents or LAR must meet this criterion.
* Participants must have a confirmed negative human immunodeficiency virus (HIV) test result within 3 months of first dose of study drug or, if unavailable, be tested by a local laboratory during the screening period.

Exclusion Criteria:

* Have CMV tissue invasive disease involving the central nervous system (CNS) or retina as assessed by the investigator at the time of screening.
* Have uncontrolled other type of infection as assessed by the investigator on the date of enrollment.
* Have a history of clinically relevant alcohol or drug abuse that may interfere with treatment compliance or assessments with the protocol as determined by the investigator.
* Be receiving valganciclovir, ganciclovir, cidofovir, foscarnet, leflunomide, letermovir, or artesunate when study treatment is initiated, or anticipated to require one of these agents during the 8-week treatment period.
* Have a known hypersensitivity to maribavir or to any excipients.
* Have severe vomiting, diarrhea, or other severe gastrointestinal (GI) illness within 24 hours prior to the first dose of study treatment or a GI absorption abnormality that would preclude administration of oral medication.
* Require mechanical ventilation or vasopressors for hemodynamic support at baseline (Visit 2/Day 1/Week 0).
* Be pregnant (or expecting to conceive) or nursing.
* Have previously completed, discontinued, or have been withdrawn from this study.
* Have received any investigational agent or device within 30 days before initiation of study treatment (includes CMV specific T-cells) or plan to receive an investigational agent or device during the study.

Previously approved agents under investigation for additional indications are not exclusionary.

* Have previously received maribavir or CMV vaccine at any time.
* Have any clinically significant medical or surgical condition that, in the investigator's opinion, could interfere with interpretation of study results, contraindicate the administration of the study treatment, or compromise the safety or well-being of the participant.
* Have severe liver disease (Child-Pugh score of >= 10).
* Have serum aspartate aminotransferase greater than (>) 5 times upper limit of normal (ULN) at screening, or serum alanine aminotransferase > 5 times ULN at screening, or total bilirubin >= 3.0 times ULN at screening (except for documented Gilbert's syndrome), as analyzed by local laboratory.
* Have positive results for HIV.
* Have active malignancy with the exception of nonmelanoma skin cancer, as determined by the investigator. Participants who experience relapse or progression of their underlying malignancy (for which HSCT or SOT was performed), as determined by the investigator, are not to be enrolled.
* Be undergoing treatment for acute or chronic hepatitis B or hepatitis C.
* Requiring ongoing treatment with or an anticipated need for treatment with a strong cytochrome P450 3A (CYP3A) inducer.
* Have a low body weight where total blood volume (TBV) required during study participation will exceed 1 percent (%) TBV per study visit or 3% TBV over a 4-week period.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  Cmax of maribavir will be evaluated.
Time to Maximum Observed Concentration (Tmax) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  Tmax of maribavir will be evaluated.
Minimum Plasma Concentration (Cmin) of Maribavir | Pre-dose; (0.5, 1.5, 3, 4, 6, and 8 hours post-dose) on Day 7 (Week 1); Pre-dose on Day 28 (Week 4); Pre-dose; (2 to 4 hours post-dose) on Day 56 (Week 8)
  Cmin of maribavir will be evaluated.
Area Under the Plasma Concentration-Time Curve Over the 1 Dosing Interval of 12 Hours at Steady State (AUC0-tau) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  AUC0-tau of maribavir will be evaluated.
Half-Life (t1/2) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  t1/2 of maribavir will be evaluated.
Terminal Elimination Rate Constant (lambdaz) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  Lambdaz of maribavir will be evaluated.
Apparent Volume of Distribution (Vz/F) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  Vz/F of maribavir will be evaluated.
Apparent Oral Clearance (CL/F) of Maribavir | Pre-dose; 0.5, 1.5, 3, 4, 6, and 8 hours post-dose on Day 7 (Week 1)
  CL/F of maribavir will be evaluated.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From start of study drug administration up to follow-up (Week 20)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily be considered related to investigational product. SAE is any untoward medical occurrence (whether considered related to investigational product or not) that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality or birth defect, or is an important medical event.

SECONDARY OUTCOMES:
Percentage of Participants With Confirmed CMV viremia Clearance at Week 8 | At Week 8
  Confirmed CMV viremia clearance is defined as plasma CMV DNA concentration below the lower limit of quantification (LLOQ) at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days at Week 8 regardless of the length of study treatment. Percentage of participants with confirmed CMV viremia clearance at Week 8 will be reported.
Percentage of Participants who Achieve Maintenance of Confirmed CMV Viremia Clearance and Symptom Control at Week 8 Through Weeks 12, 16 and 20 | At Week 8 through Weeks 12, 16, and 20
  Confirmed CMV viremia clearance is defined as plasma CMV DNA concentration below the lower LLOQ at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days regardless of the length of study treatment. CMV infection symptom control is defined as resolution or improvement of tissue invasive disease or CMV syndrome for symptomatic participants at baseline, or no new symptoms for asymptomatic participants at baseline. Percentage of participants who achieve maintenance of confirmed CMV viremia clearance and symptom control at Week 8 through Weeks 12, 16 and 20 will be reported.
Percentage of Participants With Confirmed Recurrence of CMV Viremia on Study Treatment and Off Study Treatment | Up to Week 20
  Confirmed recurrence of CMV viremia is defined as plasma CMV DNA concentration greater than or equal to (>=) LLOQ when assessed in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants with confirmed recurrence of viremia on study treatment and off study treatment will be reported.
Time to First Confirmed Viremia Clearance | Up to Week 20
  Confirmed CMV viremia clearance is defined as plasma CMV DNA concentration below the lower LLOQ when assessed at a central specialty laboratory, in 2 consecutive postbaseline samples, separated by at least 5 days. Time to first confirmed viremia clearance at any time during the study will be summarized using the Kaplan-Meier method.
Percentage of Participants With Confirmed Recurrence of CMV Viremia Treated With Alternative Anti-CMV Treatment During 12-Week Follow-up Period in Participants With Confirmed Viremia Clearance at Week 8 | From Week 8 through Week 20
  Confirmed recurrence of CMV viremia is defined as plasma CMV DNA concentration >= LLOQ when assessed in 2 consecutive plasma samples at least 5 days apart, after achieving confirmed viremia clearance. Percentage of participants with confirmed recurrence of CMV viremia treated with alternative anti-CMV treatment in the 12-Week follow-up period in participants with confirmed viremia clearance at Week 8 will be reported.
Change From Baseline in Log10 Plasma CMV Deoxyribonucleic Acid (DNA) Load | Baseline up to Week 20
  Change from baseline in log10 plasma CMV DNA on study after receiving study treatment by study week will be reported.
Number of Participants who Develop CMV Resistance to Maribavir | Up to Week 12
  CMV DNA genotyping will be performed for the UL97, UL54, UL56, and UL27 genes known to confer resistance to conventional anti-CMV therapies or Maribavir. Number of participants who developed post-baseline CMV resistance to maribavir up to Week 12 will be reported.
Summary Scores for Palatability Assessment of Maribavir | At Weeks 1, 4, and 8
  Palatability (taste, feel, smell, ease of swallowing and after-taste) is being measured using a 5-point facial hedonic scale correlated with a 100-point linear visual analogue scale (VAS) ranges from 0: very bad to 100: very good. Scores will be summarized descriptively at Weeks 1, 4 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (47):
- United States (4):
  - University of Nebraska Medical Center -985400 Nebraska Medical Center, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - Cook Children's Health Care System, Fort Worth, Texas
  - University of Texas MD Anderson Cancer Center - 1515 Holcombe Blvd, Houston, Texas
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Belgium (3):
  - Hôpital Universitaire des Enfants Reine Fabiola (HUDERF), Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent, Ghent, Oost-Vlaanderen
- Brazil (4):
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, Porto Alegre, Rio Grande do Sul
  - Hospital Do Rim E Hipertensão, São Paulo
- China (4):
  - Children's Hospital Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University - PIN, Beijing, Beijing Municipality
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences - PPDS, Tianjin, Tianjin Municipality
- France (4):
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - CHU de Grenoble Alpes - Hôpital Michallon, La Tronche, Isère
  - CHRU Nantes, Nantes, Loire-Atlantique
  - Hopital Necker, Paris
- Germany (5):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitatsklinikum Jena - Am Klinikum 1-Erlanger Allee 101, Jena, Thuringia
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Israel (4):
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center Ichilov - PPDS, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus - PPDS, Haifa
  - Hadassah Medical Center- Ein Kerem - PPDS, Petah Tikva
- Japan (5):
  - National Center for Child Health and Development, Nagoya, Aiti
  - Saitama Children's Medical Center, Isehara-Shi, Kanagawa
  - Shizuoka Children's Hospital, Aoi-ku, Shizuoka
  - Hyogo Prefectural Kobe Children's Hospital, Chiba
  - Osaka Women's and Children's Hospital, Izumi-Shi, Ôsaka
- Spain (5):
  - Hospital Sant Joan de Deu - PIN, Espluges de Llobregat, Barcelona
  - Hospital Universitario La Paz - PPDS, Horcajo de la Sierra, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Materno-Infantil, Málaga, Málaga
  - Hospital Universitario Vall d´Hebron- PPDS, Barcelona
  - Hospital Infantil Universitario Niño Jesus - PIN, Madrid
- United Kingdom (5):
  - King's College Hospital, London, Lambeth
  - Royal Manchester Children's Hospital - PIN, Manchester, Lancashire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, West Midlands
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Fisher JE, Mulieri K, Finch E, Ericson JE. Use of Maribavir for Multidrug Resistant Cytomegaloviremia in a Pediatric Oncology Patient. J Pediatr Hematol Oncol. 2024 Apr 1;46(3):e244-e247. doi: 10.1097/MPH.0000000000002841. Epub 2024 Mar 1. PMID 38447094
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/d024b354976f4ddb?idFilter=%5B%22TAK-620-2004%22%5D